CLINICAL TRIAL: NCT02931773
Title: Autonomic Cardiovascular Neuropathy in Recently Diagnosed DM2 Patients and in Pre-Diabetes Patients
Brief Title: Autonomic Cardiovascular Neuropathy in Recently Diagnosed DM2 Patients (ACNDM2)
Acronym: ACNDM2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Manuel A Sierra Beltran, Clinical Researcher, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 19677
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Dysautonomia
Keywords: Diabetes Autonomic Cardiovascular
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Probands having normal fasting glucose and having a head up tilt test with Task Force® Monitor.
  Interventions: Device: Task Force® Monitor
- Pre-Diabetes: Patients having normal fasting glucose and abnormal Oral Glucose tolerance test and having a head up tilt test with Task Force® Monitor.
  Interventions: Device: Task Force® Monitor
- Recently diagnosed Diabetic patients: Patients being diagnosed as Diabetics type in the recent five years and having a head up tilt test with Task Force® Monitor
  Interventions: Device: Task Force® Monitor

INTERVENTIONS:
Device: Task Force® Monitor — A head up tilt test carried out with a Task Force monitoring system

SUMMARY:
The investigators are studying the initial autonomic alterations in participants recently diagnosed with DM2 and in those patients classified as Pre-Diabetes, mainly focused on the baroreceptor sensitivity and on the peripheral sympathetic innervation.

DETAILED DESCRIPTION:
Until now the autonomic dysfunction in Diabetes Mellitus type 2 (DM2)has been broadly studied in long term patients. Thus, clinical features as cardiac autonomic neuropathy (CAN) and the lack of the baroreceptor reflex were widely described in patients with a long standing Diabetes. However, there hasn´t been a description of the initial autonomic imbalance in both Pre-Diabetes and recently diagnosed DM2 patients. This is the goal of the present research study, to assess the autonomic dysfunction among these sets of patients.

Yet CAN is finding mostly happening in late stages of DM2 and so the lack of Baroreceptor reflex sensitivity there are other subtle indicators of dysautonomia which hasn't been extensively analyzed. In fact, rest tachycardia and orthostatic intolerance may point to an early dysautonomia. A description of the impairment of the cardiovascular autonomic regulation is still missing. Therefore, the investigators intend to evaluate this regulation through the means of a Task Force System.

ELIGIBILITY:
Inclusion Criteria:

* patients who have not suffered Hypertension, Parkinson Diseae, Parkinsonic Syndrome, Guillain-Barré Disease, Myocardial Infarction, Obesity nor Ischemic Stroke

Exclusion Criteria:

* Those older than 55 years old, or younger than 18 years old.
* Those who have suffered Hypertension, Parkinson Diseae, Parkinsonic Syndrome, Guillain-Barré Disease, Myocardial Infarction, Obesity or Ischemic Stroke

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Those patients included as the cohorts of the GEA registry
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Sympathetic hyperactivity in recently diagnosed DM2 patients | one year
  to show that there is a cardiovascular sympathetic hyperactivity by the time of the initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manuel A Sierra-Beltrán, MD, Principal Investigator — Instituto Nacional De Cardiología "Ignacio Chávez"
Locations (1):
- Laboratio de Síncope, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
By publishing results as on as a paper on a Medical Journal